CLINICAL TRIAL: NCT01920438
Title: PEG Vs RIG: Percutaneous Endoscopic Gastrostomy Versus Radiologically Inserted Gastrostomy in Children
Brief Title: Outcome Study of Endoscopically Inserted Gastrostomy (PEG)Versus Radiologically-guided Insertion of Gastrostomy (RIG)in Children
Acronym: PEG Vs RIG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 10SG14
Record Dates: First submitted 2013-08-02; First posted 2013-08-12 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Two Interventions (PEG and RIG) Compared Against Each Other
Keywords: Percutaneous endoscopic gastrostomy,; Radiologically inserted gastrostomy,; Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEG (Experimental): Percutaneous Endoscopic Gastrostomy
  Interventions: Procedure: Percutaneous Endoscopic Gastrostomy
- RIG (Experimental): Radiologically-guided Insertion of Gastrostomy
  Interventions: Procedure: Radiologically-guided insertion of Gastrostomy

INTERVENTIONS:
Procedure: Percutaneous Endoscopic Gastrostomy — PEG
  Arms: PEG
Procedure: Radiologically-guided insertion of Gastrostomy — RIG
  Arms: RIG

SUMMARY:
A gastrostomy is a feeding tube that communicates from the skin directly into the stomach. It is a device frequently used in children that have feeding difficulties or are unable to maintain normal growth via oral feeds. The same device may be inserted in two ways: the percutaneous endoscopic method (PEG) which is guided by the use of an endoscope (flexible camera), or the radiologically inserted method (RIG) which is guided by the use of X-ray imaging. Both methods of insertion have been used in children for more than 20 years, but it is not clear which is the best method. Both methods are associated with complications, including injury to other abdominal organs and leakage leading to sepsis. There are no randomised controlled trials comparing the two techniques.

We aim to compare the outcome of both methods of gastrostomy insertion in children, with emphasis on the complication rates. We have devised a complication score with weightage assigned to each complication according to its severity.

A randomised controlled trial will be performed in children requiring a gastrostomy, 100 per group. The primary outcome will be the overall total complication rate.

ELIGIBILITY:
Inclusion Criteria:

* any child referred for gastrostomy insertion

Exclusion Criteria:

* the child has gastro-esophageal reflux and is being considered for anti-reflux surgery
* previous gastrostomy or fundoplication
* previous extensive abdominal surgery
* the child requires a concomitant major procedure on the gut or other intra- abdominal organs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-12; Primary Completion 2014-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Complication rate | 3 years
  The primary end point of the study will be the total number of complications (major and minor).

SECONDARY OUTCOMES:
1. major complication rate : complications requiring surgery | 3 years
  Colonic injury or gastro-colic fistula or other visceral injury, peritonitis requiring surgery, intestinal obstruction requiring surgery, major gastrointestinal bleed, other complications requiring surgery
2. minor complication rate : complications not requiring surgery | 3 years
  Infection requiring systemic antibiotics, delay more than 48 hours in establishing feeds, granulation, wound site discharge, tube-related problems (migration, dislodgement, leakage, breakage), other minor
3.complication score | 3 years
  This is a score devised with weighting assigned to each complication depending on the severity of the complication.The score was devised in a consensus meeting attended by experts in the field (paediatric surgeons, interventional radiologists, junior doctors and nurses.
4.technical failure | 3 yaers
  These are the number of PEG or RIG that are unsuccessful and require conversion to open surgical gastrostomy or laparoscopic gastrostomy.
5.difficulty of procedure | 3 years
  Assessed by the operator as : 1) easy, 2) slightly difficult (but does not warrant conversion), 3) difficult (warrants conversion)
6.cost of hospital treatment | 3 years
7.mortality | 3 years
8.cause of death | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Joe I Curry, MBBS,FRCS(Eng),FRCS(Paed Surg), Study Chair — Great Ormond Street Hospital Great Ormond Street, London, WC1N 3JHLondon
Locations (1):
- Great Ormond Street Hospital, London, United Kingdom

REFERENCES:
- [Background] Nah SA, Narayanaswamy B, Eaton S, Coppi PD, Kiely EM, Curry JI, Drake DP, Barnacle AM, Roebuck DJ, Pierro A. Gastrostomy insertion in children: percutaneous endoscopic or percutaneous image-guided? J Pediatr Surg. 2010 Jun;45(6):1153-8. doi: 10.1016/j.jpedsurg.2010.02.081. PMID 20620311
- [Derived] Singh RR, Nah SA, Roebuck DJ, Eaton S, Pierro A, Curry JI; PEG-RIG trial collaborators. Double-blind randomized clinical trial of percutaneous endoscopic gastrostomy versus radiologically inserted gastrostomy in children. Br J Surg. 2017 Nov;104(12):1620-1627. doi: 10.1002/bjs.10687. Epub 2017 Sep 20. PMID 28940403